CLINICAL TRIAL: NCT02649361
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Trial to Compare the Efficacy and Safety of Anlotinib Versus Placebo in Patients With Esophageal Squamous Cell Carcinoma(ALTER1102)
Brief Title: Study of Anlotinib in Patients With Esophageal Squamous Cell Carcinoma (ALTER1102)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTN-11-II
Record Dates: First submitted 2016-01-06; First posted 2016-01-07 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Anlotinib
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — anlotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anlotinib (Experimental): Anlotinib QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Anlotinib
- Placebo (Placebo Comparator): Placebo QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anlotinib — Anlotinib p.o. qd
  Arms: Anlotinib
Drug: Placebo — Placebo p.o. qd
  Arms: Placebo

SUMMARY:
To compare the effects and safety of Anlotinib with placebo in patients with esophageal squamous cell carcinoma(ESCC).

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of esophageal squamous cell carcinoma；
* Advanced esophageal squamous cell carcinoma with distant metastasis(Stage IV),at least one measurable lesion (by RECIST1.1)
* Patients who at least have failed to a platinum-based chemotherapy treatment or chemotherapy containing paclitaxel.

Note: (1) Each line treatment refers to treatment duration at least one cycle using monotherapy or drug combination; (2)Adjuvant chemotherapy or neoadjuvant chemoradiation is permitted before the study (if disease recurred during adjuvant chemotherapy/neoadjuvant chemoradiation or recurred within 6 months after stopping treatment, adjuvant chemotherapy/neoadjuvant chemoradiation can be considered as first line systemic chemotherapy;

* 18-75 years,ECOG PS:0-2,Life expectancy of more than 3 months
* 4 weeks or more from the last cytotoxic therapy, radiation therapy or surgery
* Main organs function is normal
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped
* Patients should participate in the study voluntarily and sign informed consent

Exclusion Criteria:

* Patients whose primary lesion with active bleeding within 2 months
* Primary lesion not resected and has not shrinked after radiation therapy
* Patients who have been failure with anti-tumor angiogenesis drug treatment
* Patients with factors that could affect oral medication (such as dysphagia，chronic diarrhea, intestinal obstruction etc.)
* Brain metastases patients with symptoms or symptoms controlled < 3 months
* Patients with any severe and/or unable to control diseases，including：

  1. Blood pressure unable to be controlled ideally(systolic pressure≥150 mmHg，diastolic pressure≥100 mmHg);
  2. Patients with Grade 1 or higher myocardial ischemia, myocardial infarction or malignant arrhythmias(including QT≥480ms) and patients with Grade 1 or higher congestive heart failure (NYHA Classification);
  3. Patients with active or unable to control serious infections;
  4. Patients with cirrhosis, decompensated liver disease, or active hepatitis;
  5. Patients with poorly controlled diabetes (fasting blood glucose(FBG)>10mmol/L)
  6. Urine protein ≥ ++，and 24-hour urinary protein excretion>1.0 g confirmed
* Patients with non-healing wounds or fractures
* Patients with any CTC AE Grade 1 or higher bleeding events occurred in the lungs or any CTC AE Grade 2 or higher bleeding events occurred within 4 weeks prior to assignment;Patients with any physical signs of bleeding diathesis or receiving thrombolysis and anticoagulation
* Patients with arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism
* Patients with drug abuse history and unable to get rid of or Patients with mental disorders
* Imaging showed tumors have involved important blood vessels or by investigators determine likely during the follow-up study and cause fatal hemorrhage
* Patients participated in other anticancer drug clinical trials within 4 weeks
* History of immunodeficiency
* Patients with concomitant diseases which could seriously endanger their own safety or could affect completion of the study according to investigators' judgment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2016-01; Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

PRIMARY OUTCOMES:
Progress free survival (PFS) | From randomization，each 42 days up to PD or death(up to 24 months)

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization until death (up to 24 months)
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Harbin medical university affiliated tumor hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Shandong Cancer Hospital, Jinan, Shandong
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xian Jiaotong University, Xian, Shanxi
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality
  - Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang J, Xiao J, Fang W, Lu P, Fan Q, Shu Y, Feng J, Zhang S, Ba Y, Zhao Y, Liu Y, Bai C, Bai Y, Tang Y, Song Y, He J. Anlotinib for previously treated advanced or metastatic esophageal squamous cell carcinoma: A double-blind randomized phase 2 trial. Cancer Med. 2021 Mar;10(5):1681-1689. doi: 10.1002/cam4.3771. Epub 2021 Feb 14. PMID 33586360